CLINICAL TRIAL: NCT04552015
Title: Pilot Study for Development of Microneedles for Diagnosis of Latent Tuberculosis Infection
Brief Title: Microneedles for Diagnosis of LTBI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: There is a problem with the investigational product
Sponsor: The HIV Netherlands Australia Thailand Research Collaboration (Other)
Collaborators: National Nanotechnology Center (NANOTEC), The National Science and Technology Development Agency (NSTDA) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HIV-NAT 276
Record Dates: First submitted 2020-09-10; First posted 2020-09-17 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Latent Tuberculosis
MeSH Terms: conditions — Latent Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- volunteers (Other): two different types of diagnostic tools (TST vs microneedle) will be used to screen for latent TB infection
  Interventions: Diagnostic Test: TST vs PPD microneedle test

INTERVENTIONS:
Diagnostic Test: TST vs PPD microneedle test — TST vs First patch: 800 um in length, PPD1 formulation; Second patch: 1,500 um in length, PPD1 formulation; Third patch: 800 um in length, PPD2 formulation; and Fourth patch: 1,500 um in length, PPD2 formulation

SUMMARY:
This study will evaluate new technique, microneedle, to detect latent tuberculosis (TB) in healthy volunteers

DETAILED DESCRIPTION:
The cross-sectional study to investigate the effect of microneedle formulations and lengths of Tuberculin PPD microneedles on the delayed-type hypersensitivity response in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Sex : Male and Female
2. Age : 20-60 years
3. TB contacts or those at risk of TB e.g. health-care workers
4. HIV-negative healthy individuals

Exclusion Criteria:

1. Presence of an acute infection, as determined by investigators
2. Receiving immunosuppression drugs e.g. steroids
3. Having autoimmune diseases e.g. SLE (Systemic Lupus Erythematous)
4. Being pregnant or breastfeeding

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2021-04-08 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
size of induration at 48 hours post-PPD injection | 48 hours
  Monitoring the response of delayed-type hypersensitivity on the skin by comparing TST to microneedle tests

CONTACTS AND LOCATIONS:
Overall Officials: Sivaporn Gatechompol, MD, Principal Investigator — The HIV Netherlands Australia Thailand Research Collaboration; Jeerapond Leelawattanachai, PhD, Principal Investigator — King Chulalongkorn Memorial Hospital; Saradee Warit, PhD, Principal Investigator — King Chulalongkorn Memorial Hospital
Locations (1):
- Faculty of Medicine, Chulalongkorn University, Bangkok, Thailand